CLINICAL TRIAL: NCT03350620
Title: A 3-Arm Randomized, Double-Masked, Placebo-Controlled, Phase 3 Study of NVK-002 in Children With Myopia
Brief Title: CHAMP: Study of NVK-002 in Children With Myopia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vyluma, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Organization: Nevakar, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP-NVK002-0001; 2018-001077-24 (EudraCT Number)
Record Dates: First submitted 2017-11-16; First posted 2017-11-22 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-10

CONDITIONS: Myopia
Keywords: child, myopia, nearsightedness
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: This will be a 3-arm randomized, multicenter, double-masked, placebo-controlled study conducted in 2 stages. Stage 1 is to assess the primary and secondary endpoints. Stage 2 is an extension stage for exploratory endpoints.
  Stage 1 is a safety and efficacy phase of 3 years in duration, during which subjects will be allocated to 1 of 3 study medications.
  Stage 2 is a randomized cross-over phase of 1 year in duration, during which subjects will be re-randomized to receive 1 of the 3 study medications with subjects initially randomized to Vehicle only eligible for randomization to low or high dose NVK-002.
Who Masked: Participant, Investigator
Masking Description: If subjects meet eligibility criteria at the Screening/Baseline visit (Day 0), subjects will be randomly assigned to masked study medication.
  The study will be double masked. The study medication will be provided in identical-appearing laminated pouches with no labeling indicating the identity of the study group or the contents of the ampules. The laminated pouches will contain identical-appearing ampules. Study subjects and study management personnel will be masked to the identity of treatment until after the final database lock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NVK-002 Concentration 1 (Experimental): Stage 1: Subjects will be randomized to NVK-002 Concentration 1
  Stage 2: Subjects will be re-randomized to one of the three treatment arms.
  Interventions: Drug: NVK-002 Concentration 1
- NVK-002 Concentration 2 (Experimental): Stage 1: Subjects will be randomized to NVK-002 Concentration 2
  Stage 2: Subjects will be re-randomized to one of the three treatment arms.
  Interventions: Drug: NVK-002 Concentration 2
- Vehicle (Placebo) (Placebo Comparator): Stage 1: Subjects will be randomized to Vehicle (Placebo)
  Stage 2: Subjects will be re-randomized to one of the two experimental NVK-002 treatment arms
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NVK-002 Concentration 1 — Study medication will be administered, once daily (QD)
  Other Names: NVK-002 Conc 1
  Arms: NVK-002 Concentration 1
Drug: NVK-002 Concentration 2 — Study medication will be administered, once daily (QD)
  Other Names: NVK-002 Conc 2
  Arms: NVK-002 Concentration 2
Drug: Placebo — Vehicle (placebo) will be administered, once daily (QD)
  Other Names: Vehicle
  Arms: Vehicle (Placebo)

SUMMARY:
Stage 1: To evaluate the safety and efficacy of 2 concentrations of NVK-002 compared to Vehicle (placebo) for slowing the progression of myopia in children over a 3 year treatment period.

Stage 2: To observe safety and efficacy in subjects re-randomized to one (1) year of treatment with NVK-002 or Vehicle following 3 years of treatment in children with progressive myopia.

DETAILED DESCRIPTION:
This will be a 3-arm randomized, multicenter, double-masked, placebo-controlled study conducted in 2 stages.

Stage 1 is a safety and efficacy phase of 3 years in duration, during which subjects will be allocated to 1 of 3 study medications.

Stage 2 is a randomized follow-up phase of 1 year in duration, during which subjects will be re-randomized to receive 1 of the 3 study medications, with subjects initially randomized to Vehicle only eligible for randomization to low or high-dose NVK-002.

Treatment arms are:

* NVK-002 low dose concentration
* NVK-002 high dose concentration
* Vehicle (placebo)

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 3 to ≤ 17.0 years.
2. Myopia SER of at least -0.50 D and no worse than -6.00 D myopia in each eye as measured by cycloplegic autorefraction.

Exclusion Criteria:

1. If present, astigmatism more than -1.50 D in either eye.
2. Current or history of amblyopia or strabismus.
3. History of any disease or syndrome that predisposes the subject to severe myopia (e.g., Marfan syndrome, Stickler syndrome, retinopathy of prematurity).
4. History in either eye of abnormal ocular refractive anatomy (e.g., keratoconus, lenticonus, spherophakia).
5. Serious systemic illness that, in the Investigator's opinion, would render the subject ineligible.
6. Chronic use (more than 3 days per week) of any topical ophthalmic medications (prescribed or over the-counter) other than the assigned study medication.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 670 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Houman Hemmati, MD, Study Director — Nevakar, Inc.
Locations (26):
- United States (20):
  - Site #009, Tucson, Arizona
  - Site #015, Berkeley, California
  - Site #003, Fullerton, California
  - Site #016, San Diego, California
  - Site #005, Danbury, Connecticut
  - Site #004, Maitland, Florida
  - Site #024, Peoria, Illinois
  - Site #006, Boston, Massachusetts
  - Site #014, St Louis, Missouri
  - Site #002, New York, New York
  - Site #013, Raleigh, North Carolina
  - Site #001, Columbus, Ohio
  - Site #018, Forest Grove, Oregon
  - Site #011, Elkins Park, Pennsylvania
  - Site #017, Lancaster, Pennsylvania
  - Site #008, Memphis, Tennessee
  - Site #007, San Antonio, Texas
  - Site #012, Kirkland, Washington
  - Site #020, Spokane, Washington
  - Site #021, Madison, Wisconsin
- Site #104, Budapest, Hungary
- Site #101, Dublin, Ireland
- Site # 105, Rotterdam, Netherlands
- Site #107, Barcelona, Spain
- United Kingdom (2):
  - Site #103, Coleraine
  - Site #106, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zadnik K, Schulman E, Flitcroft I, Fogt JS, Blumenfeld LC, Fong TM, Lang E, Hemmati HD, Chandler SP; CHAMP Trial Group Investigators. Efficacy and Safety of 0.01% and 0.02% Atropine for the Treatment of Pediatric Myopia Progression Over 3 Years: A Randomized Clinical Trial. JAMA Ophthalmol. 2023 Oct 1;141(10):990-999. doi: 10.1001/jamaophthalmol.2023.2097. PMID 37261839

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled subjects who did not meet the inclusion criteria or met the exclusion criteria were not randomized.
Groups:
- NVK-002 Concentration 1: Stage 1: Subjects will be randomized to NVK-002 Concentration 1
  Stage 2: Subjects will be re-randomized to one of the three treatment arms.
  NVK-002 Concentration 1: Study medication will be administered, once daily (QD)
- NVK-002 Concentration 2: Stage 1: Subjects will be randomized to NVK-002 Concentration 2
  Stage 2: Subjects will be re-randomized to one of the three treatment arms.
  NVK-002 Concentration 2: Study medication will be administered, once daily (QD)
- Vehicle (Placebo): Stage 1: Subjects will be randomized to Vehicle (Placebo)
  Stage 2: Subjects will be re-randomized to one of the two experimental NVK-002 treatment arms
  Placebo: Vehicle (placebo) will be administered, once daily (QD)
Period: Stage 1
Arm/Group | NVK-002 Concentration 1 | NVK-002 Concentration 2 | Vehicle (Placebo)
Started | 164 | 247 | 165 (3 participants were assigned to placebo but did not take at least 1 dose of assigned treatment. hence N=165 for ITT in efficacy assessment and N=162 for the safety set used in TEAE reporting)
Completed | 127 | 207 | 143
Not Completed | 37 | 40 | 22
Period: Stage 2
Arm/Group | NVK-002 Concentration 1 | NVK-002 Concentration 2 | Vehicle (Placebo)
Started (Per Statistical Analysis Plan, Stage 2 outcomes are all exploratory and tertiary outcomes.) | 159 (Stage 2 concentration 1 is combined from 3 parallel groups: stage 1 placebo to stage 2 concentration 1 (N=62); stage 1 concentration 1 to stage 2 concentration 1 (N=38); stage 1 concentration 2 to stage 2 concentration 1 (N=59).) | 162 (Stage 2 concentration 2 is combined from 3 parallel groups: stage 1 placebo to stage 2 concentration 2 (N=60); stage 1 concentration 1 to stage 2 concentration 2 (N=39); stage 1 concentration 2 to stage 2 concentration 2 (N=63).) | 99 (Stage 2 Placebo is combined from 2 parallel groups: stage 1 concentration 1 to stage 2 Placebo (N=39); stage 1 concentration 2 to stage 2 Placebo (N=60).)
Completed | 156 | 153 | 96
Not Completed | 3 | 9 | 3
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — unable to visit (1); used prohibited concomitant medication / withdrew consent (4); relocation (1). | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVK-002 Concentration 1 | NVK-002 Concentration 2 | Vehicle (Placebo) | Total
Number analyzed (Participants) | 164 | 247 | 165 | 576
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (2.1) | 9.0 (2.1) | 8.8 (1.8) | 8.9 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 136 | 94 | 315
  Male | 79 | 111 | 71 | 261
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 1 | 7
  Asian | 29 | 54 | 26 | 109
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 3 | 4
  Black or African American | 23 | 31 | 27 | 81
  White | 84 | 132 | 93 | 309
  More than one race | 15 | 7 | 8 | 30
  Unknown or Not Reported | 9 | 20 | 7 | 36
Region of Enrollment [Number; unit: participants]
  Europe | 34 | 48 | 29 | 111
  United States | 130 | 199 | 136 | 465
SER [Median (Inter-Quartile Range); unit: Diopter] | -2.25 [-5.87 to -0.50] | -2.33 [-5.87 to -0.50] | -2.41 [-5.90 to -0.50] | -2.33 [-5.90 to -0.50]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects' Eyes That Show < 0.50 D Myopia Progression (SER, Spherical Equivalent Refraction) at the Month 36 Visit
Description: Number of subjects' eyes that show < 0.50 D myopia progression (SER, spherical equivalent refraction) at the Month 36 visit.
Time Frame: 36 Months
Population: ITT
Measure: Number; unit: participants' eyes
Units Other Than Participants: participants' eyes
Arm/Group | NVK-002 Concentration 1 | NVK-002 Concentration 2 | Vehicle (Placebo)
Number analyzed (Participants) | 164 | 247 | 165
Number analyzed (participants' eyes) | 328 | 494 | 330
participants' eyes | 79 | 106 | 61

2. Secondary Outcome: Change From Baseline in SER (Spherical Equivalent Refraction)
Description: Change from baseline in SER (spherical equivalent refraction).
Time Frame: Month 36
Population: ITT
Measure: Median (Inter-Quartile Range); unit: Diopter
Units Other Than Participants: Participants' eyes
Arm/Group | NVK-002 Concentration 1 | NVK-002 Concentration 2 | Vehicle (Placebo)
Number analyzed (Participants) | 164 | 247 | 165
Number analyzed (Participants' eyes) | 328 | 494 | 330
Diopter | -0.85 [-3.28 to 1.22] | -1.02 [-3.94 to 0.89] | -1.10 [-4.44 to 3.60]

ADVERSE EVENTS:
Time Frame: 3 years (Stage 1) and 1 year (Stage 2)
Description: Treatment-emergent adverse events (TEAEs) are defined as any new or worsening of existing adverse events that occur or worsen between the first dose date of a specific stage and the last dose date of the same stage.
  All-cause mortality, serious AE and other AE reporting are based on the Safety Set. The Safety Set (SS) will include all subjects who were administered at least one dose of study medication in Stage 1 or Stage 2.
Groups:
- Stage 1: NVK-002 Concentration 1: Stage 1: Subjects randomized to NVK-002 Concentration 1
  NVK-002 Concentration 1: Study medication will be administered, once daily (QD)
- Stage 1: NVK-002 Concentration 2: Stage 1: Subjects randomized to NVK-002 Concentration 2
  NVK-002 Concentration 2: Study medication will be administered, once daily (QD)
- Stage 1: Vehicle (Placebo): Stage 1: Subjects randomized to Vehicle (Placebo)
  Placebo: Vehicle (placebo) will be administered, once daily (QD).
  Note: N=162 for the safety set (see comment in participant flow)
- Stage 2: NVK-002 Concentration 1: Stage 2: Subjects randomized to NVK-002 Concentration 1 include those from Stage 1 NVK-002 concentration, Stage 1 NVK-002 concentration 2 and Stage 1 Vehicle (Placebo).
- Stage 2: NVK-002 Concentration 2: Stage 2: Subjects randomized to NVK-002 Concentration 2 include those from Stage 1 NVK-002 concentration 1, NVK-002 concentration 2, and Stage 1 Vehicle (Placebo).
- Stage 2: Vehicle (Placebo): Stage 2: Subjects randomized to Vehicle (Placebo) include those from Stage 1 NVK-002 concentration 1 and Stage 1 NVK-002 concentration 2.
Arm/Group | Stage 1: NVK-002 Concentration 1 | Stage 1: NVK-002 Concentration 2 | Stage 1: Vehicle (Placebo) | Stage 2: NVK-002 Concentration 1 | Stage 2: NVK-002 Concentration 2 | Stage 2: Vehicle (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/164 | 0/247 | 0/162 | 0/159 | 0/162 | 0/99
Serious Adverse Events (participants affected / at risk) | 1/164 | 8/247 | 4/162 | 3/159 | 2/162 | 2/99
Other Adverse Events (participants affected / at risk) | 56/164 | 92/247 | 75/162 | 43/159 | 29/162 | 17/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: NVK-002 Concentration 1 (N=164) | Stage 1: NVK-002 Concentration 2 (N=247) | Stage 1: Vehicle (Placebo) (N=162) | Stage 2: NVK-002 Concentration 1 (N=159) | Stage 2: NVK-002 Concentration 2 (N=162) | Stage 2: Vehicle (Placebo) (N=99)
Appendicitis (Infections and infestations) | 0 | 2 | 2 | 1 | 0 | 0
COVIV-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Parainfluenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anal fisuure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
seizure (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Disruptive mood dysregulation disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mania (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ankle fracture (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: NVK-002 Concentration 1 (N=164) | Stage 1: NVK-002 Concentration 2 (N=247) | Stage 1: Vehicle (Placebo) (N=162) | Stage 2: NVK-002 Concentration 1 (N=159) | Stage 2: NVK-002 Concentration 2 (N=162) | Stage 2: Vehicle (Placebo) (N=99)
nasopharyngitis (Infections and infestations) | 17 | 30 | 22 | 14 | 5 | 6
COVID-19 (Infections and infestations) | 9 | 27 | 18 | 14 | 13 | 8
influenza (Infections and infestations) | 6 | 8 | 12 | 4 | 2 | 2
hordeolum (Infections and infestations) | 3 | 10 | 11 | 2 | 2 | 1
ocular hyperemia (Eye disorders) | 4 | 8 | 10 | 0 | 0 | 0
headache (Nervous system disorders) | 14 | 23 | 14 | 5 | 2 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 9 | 2 | 2 | 0
seasonal allergy (Immune system disorders) | 12 | 14 | 9 | 5 | 4 | 1
pyrexia (General disorders) | 8 | 21 | 6 | 3 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT03350620/Prot_001.pdf
  • Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT03350620/SAP_000.pdf